CLINICAL TRIAL: NCT03540498
Title: Oral Colonization by Lactobacillus Brevis KABP 052 (CECT 7480) and Lactobacillus Plantarum KABP 051 (CECT 7481): A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Study of Colonization of Strains L.Plantarum and L.Brevis in the Product AB-DENTALAC Chewing Gum
Acronym: AB-GUM-2016
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Collaborators: Clínica Odontológica Nart en Barcelona (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB-GUM-2016
Record Dates: First submitted 2018-05-07; First posted 2018-05-30 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Periodontal Disease
Keywords: Oral health; Probiotics; L. plantarum; L. brevis; Periodontics; Dental plaque
MeSH Terms: conditions — Periodontal Diseases; Dental Plaque | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: The study will follow a randomized, double-blind, split-mouth, placebo-controlled design with two parallel prospective follow-up groups for the evaluation of two different posology models (with or without previous professional oral cleaning).
Who Masked: Participant, Investigator
Masking Description: Once the patients have been selected according to the inclusion / exclusion criteria detailed below, they will be included in one of the treatment groups (control / study) in a random and random manner. The list of randomization and the labeling of the products will be carried out by independent personnel to the research team to ensure double blindness of the trial. The production of the probiotic products and control will be carried out in both cases in white boxes without any type of identification or difference between them.
  The randomization will be made from an online software available at www.randomization.com. From the list of randomization generated by this software, the different products will be labeled with the patient number and the test code. The team of researchers will not have access to the randomization list. In this way, a correct randomization and double-blind trial is guaranteed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): The volunteers will follow the assigned treatment for 6 weeks (PROBIOTICS_AB-DENTALAC CHEWING GUM. Orally) , which will consist of the consumption of 2 chewing gums a day. The chewing gum should be chewed for at least 15-20 minutes at least 1 hour after the consumption of food. For at least 1 hour after the consumption of chewing gum, volunteers will not be able to consume food, drink (except water) or clean their teeth. Adherence to the treatment will be made by returning the empty containers after 6 weeks.
  Interventions: Dietary Supplement: AB-DENTALAC [Probiotics (study)]
- Control (Placebo Comparator): The volunteers will follow the assigned treatment for 6 weeks (PLACEBOS CHEWING GUM. Orally) , which will consist of the consumption of 2 chewing gums a day. The chewing gum should be chewed for at least 15-20 minutes at least 1 hour after the consumption of food. For at least 1 hour after the consumption of chewing gum, volunteers will not be able to consume food, drink (except water) or clean their teeth. Adherence to the treatment will be made by returning the empty containers.
  Interventions: Dietary Supplement: Placebo (control)

INTERVENTIONS:
Dietary Supplement: AB-DENTALAC [Probiotics (study)] — Treatment for 6 weeks, which will consist of the consumption of a chewing gum AB-DENTALAC with 100mg L.plantarum + L.brevis Probiotics blend (5E+8 CFU each at the end of shelf life), b.i.d (morning and evening).
  Arms: Probiotics
Dietary Supplement: Placebo (control) — Treatment for 6 weeks, which will consist of the consumption of a chewing gum placebo, without probiotics strains, b.i.d (morning and evening).
  Arms: Control

SUMMARY:
Study will follow a randomized, double-blind, placebo-controlled design with two groups in parallel,N of 40 patients in 6 weeks of follow up for the evaluation of two different posology models (daily consumption of probiotic gum, with or without previous professional oral cleaning). Probiotics have recently been used to combat oral diseases (plaque control, caries, halitosis, etc.), as a non-invasive natural therapy.

DETAILED DESCRIPTION:
The study will follow a randomized, double-blind, placebo-controlled design with two groups in parallel, for the evaluation of two different posology models (daily consumption of probiotic gum, with or without previous professional oral cleaning). Probiotics have recently been used to combat oral diseases (plaque control, caries, halitosis, etc.), as a non-invasive natural therapy.

The aim of this study is to assess whether the daily consumption of AB-DENTALAC gum allows the colonization of strains L.plantarum KABP051 (CECT7481) and L.brevis KABP052 (CECT7480) in the oral microbiota, and to confirm the absence of side effects, with the following setup:

1. Number of patients to be randomized:40
2. Number of visits per patient: 2

The study will determine the index of plaque and gingival index as a measure of oral health. The presence of Lactobacillus in the samples collected by qPCR will also be quantified.

The patient will benefit from a buccal revision and control by a periodontist for 6 weeks. It will also help subsequent patients to obtain a better treatment (if the results are significant). No harm is expected to participate, it is a minimal risk study, with non-invasive exploratory tests and a product suitable for human consumption and marketed in Europe since 2012.

The potential patients to participate in the study will be healthy patients, so if they do not wish to participate they will not need alternative treatment. The objective of the study is to see if the probiotic is able to colonize the mouth in healthy patients, it is not a study to demonstrate the effectiveness of the product.

If there is any serious adverse effect (something totally unexpected being a product with probiotic strains QPS), the patient will be advised to stop taking the product immediately. It is not anticipated that the use of any additional treatment is necessary.

The promoter will provide all the necessary material for the study: 60 cases of placebo chewing gum, 60 cases of probiotic chewing gum, and cleaning material (toothbrush and fluoridated toothpaste) for all patients.

Statistical analysis of bacterial colonization will be performed using Student's T with logarithmic transformation of data if required, considering a two-tailed P <0.05 as significance cut-off.

ELIGIBILITY:
Inclusion Criteria:

* Women and men between 18-55 years.
* Capacity to understand the procedures and implications of the study.
* Gingival Index <1,5 (Löe and Silness, Acta Odontol Scand. 1963. 21:533-51)
* Plaque Index <2,0 (Löe and Silness, Acta Odontol Scand. 1963. 21:533-51)
* Periodontal pocket depth <5 mm

Exclusion Criteria:

* Less than 20 natural teeth
* More than 2 untreated caries at the time of enrollment
* Current orthodontic or periodontal treatment
* Hypersensitivity or allergy to any of the ingredients of the experimental product
* Consumption of antibiotics in the 8 weeks prior to treatment
* Use of probiotics designed to improve oral health, or having consumed them during the 8 weeks prior to the study
* Consumption of any type of probiotic during the 4 weeks prior to the study
* Usual consumption of clorhexidine or other mouthwashes with bactericidal active ingredients during the 30 days before the start of the study
* Pregnant or lactating women
* Participants with chronic diseases (eg, diabetes, kidney problems, cancer) or under chronic treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Probiotic colonization of the oral cavity (qPCR) | Change from Baseline assessed 6 weeks after study entry
  Quantification of L. brevis and L. plantarum by species-specific qPCR in pooled samples of saliva, dental plaque (from the CPI subset) and lingual plaque

SECONDARY OUTCOMES:
Progression of PII | Change from Baseline assessed 6 weeks after study entry
  Plaque Index (PlI; Silness and Löe 1964) in the CPI teeth subset, as recorded at the first visit and at the end of the study by the dentist.
Progression of GI | Change from Baseline assessed 6 weeks after study entry
  Gingival Index (GI; Löe and Silness 1963) in the CPI teeth subset, as recorded at the first visit and at the end of the study by the dentist.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Espadaler Mazo, PhD, Study Chair — AB Biotics, SA; Jose Nart Molina, DMD, Principal Investigator — Clínica Odontológica Nart en Barcelona

REFERENCES:
- [Derived] Nart J, Jimenez-Garrido S, Ramirez-Sebastia A, Asto E, Buj D, Huedo P, Espadaler J. Oral colonization by Levilactobacillus brevis KABPTM-052 and Lactiplantibacillus plantarum KABPTM-051: A Randomized, Double-Blinded, Placebo-Controlled Trial (Pilot Study). J Clin Exp Dent. 2021 May 1;13(5):e433-e439. doi: 10.4317/jced.57771. eCollection 2021 May. PMID 33981389